CLINICAL TRIAL: NCT03059641
Title: Mutation Profile Detection, Therapeutic Resistance and Clonal Evolution Assessed With Liquid Biopsy of Advanced NSCLC Patients in China
Brief Title: Therapeutic ResistAnce and Clonal Evolution Assessed With Liquid Biopsy of NSCLC Patients in China
Status: Completed | Type: Observational
Sponsor: Geneplus-Beijing Co. Ltd. (Industry)
Collaborators: Shanghai Chest Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TRACELib-NSCLC
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Lung Neoplasms; Lung Cancer, Nonsmall Cell; Adenocarcinoma of Lung; Squamous Cell Lung Cancer
Keywords: Next Generation Sequencing (NGS); Tyrosine Kinase Inhibitor (TKI); liquid biopsy; EGFR Gene mutation
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood (including plasma, white cells), tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the concordance of sensitizing mutations detected between paired plasma and tissue samples; the correlation between the clonal status of sensitizing mutations and targeted therapy response; and the prognostic impact of the relative abundance of sensitizing / resistance mutations.

DETAILED DESCRIPTION:
In the study, 500 advanced NSCLC patients will be recruited. All the patients will receive biopsy genotype assay and circultating tumor DNA (ctDNA) liquid biopsy. Patients who carry actionable EGFR mutation, ROS1 fusion, ALK fusion or MET exon 14 skipping mutation will receive TKI treatment according to guidelines. During the TKI treatment, every patients will take liquid biopsy assay to monitor the mutation status. The study will be ended when all the patients had a progressive disease (PD) in their targeted lesion.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Newly diagnosed and histological or cytological confirmed stage IIIB-IV lung adenocarcinoma or non-smoking squamous cell carcinoma patients according to the AJCC staging system. The stage IV lung cancer and brain metastasis can be diagnosed by imaging and enhanced CT respectively
* ECOG performance status 0-2 with expected more than 6 months of survival time
* Willingness to comply with required protocols and give permission to use the data for clinical research and products development

Exclusion Criteria:

* Patients have other primary cancers
* Patients have symptomatic brain metastasis, complications that are associated with brain metastasis or cognitive disorders
* Patients failed in either plasma or tissue sample QC

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: treatment naïve Stage IIIB or Stage IV NSCLC patients, adenocarcinoma or squamous cell carcinoma without smoking history
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
The mutation pattern of untreated advanced NSCLC and evolution of ctDNA mutation profile during TKI treatment. | 2 years

SECONDARY OUTCOMES:
The concordance of gene mutation pattern between liquid biopsy and tissue biopsy. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD, Principal Investigator — Shanghai Chest Hospital
Locations (14):
- China (14):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - First Hospital of Jilin University, Changchun
  - Sir Run Run Shaw Hospital, Zhejiang University School of medicine, Hangzhou
  - The First Hospital of Zhejiang Province, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - Jiangsu Jiangyin People's Hospital, Jiangyin
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Ningbo No.2 Hospital, Ningbo
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Shanghai East Hospital, Shanghai
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Affiliated Hospital, Jiangnan University, Wuxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ai X, Cui J, Zhang J, Chen R, Lin W, Xie C, Liu A, Zhang J, Yang W, Hu X, Hu X, Zhao Q, Rao C, Zang YS, Ning R, Li P, Chang L, Yi X, Lu S. Clonal Architecture of EGFR Mutation Predicts the Efficacy of EGFR-Tyrosine Kinase Inhibitors in Advanced NSCLC: A Prospective Multicenter Study (NCT03059641). Clin Cancer Res. 2021 Feb 1;27(3):704-712. doi: 10.1158/1078-0432.CCR-20-3063. Epub 2020 Nov 13. PMID 33188140